CLINICAL TRIAL: NCT03171831
Title: Haploidentical Hematopoietic Stem Cell Transplantation for Patients With Thalassemia Major
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yongrong Lai, Director of the Hematology Department, First Affiliated Hospital of Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Guangxi-Haplo-HSCT-2016
Record Dates: First submitted 2017-04-18; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — Busulfan; Cyclophosphamide; fludarabine; Influenza Vaccines; Mycophenolic Acid; Tacrolimus; Methotrexate; thymoglobulin; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Haploidentical HSCT (Experimental): Procedure: Haploidentical hematopoietic stem cell transplantation from a related donor (partially matched sibling, father or mother).
  Conditioning: Busulfan （4 mg/kg/day,4 days） + Cyclophosphamide （50 mg/kg/day,4 days）+ Fludarabine （50 mg/m2/day,3 days）
  GVHD Prophylaxis：Mycophenolate mofetil（0.25g/day）+ Tacrolimus（0.03mg/kg/day）+ Methotrexate（15mg/m2 on day +1,10mg/m2 on day +3,+6,+11）+ Thymoglobulin（2.5 mg/kg/day,4 days）+Basiliximab（10mg on day 0 and +4）
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Methotrexate; Drug: Thymoglobulin; Drug: Basiliximab

INTERVENTIONS:
Drug: Busulfan — Busulfan（4 mg/kg/day,4 days）
  Other Names: Bu
Drug: Cyclophosphamide — Cyclophosphamide（50 mg/kg/day,4 days）
  Other Names: Cy
Drug: Fludarabine — Fludarabine（50 mg/m2/day,3 days）
  Other Names: Flu
Drug: Mycophenolate mofetil — Mycophenolate mofetil（0.25g/day）
  Other Names: MMF
Drug: Tacrolimus — Tacrolimus（0.03mg/kg/day）
  Other Names: FK506
Drug: Methotrexate — Methotrexate（15mg/m2 on day +1,10mg/m2 on day +3,+6,+11）
  Other Names: MTX
Drug: Thymoglobulin — Thymoglobulin（2.5 mg/kg/day,4 days）
  Other Names: ATG
Drug: Basiliximab — Basiliximab（10mg on day 0 and +4）
  Other Names: Simulect

SUMMARY:
The purpose of the study is to assess the safety and efficacy of haploidentical hematopoietic stem cell transplantation for patients with thalassemia major.

DETAILED DESCRIPTION:
The only curative therapy for thalassemia major remains the replacement of the defective erythropoiesis by allogeneic hematopoietic stem cell transplantation(HSCT). However, this option is unavailable to many patients as a result of a lack of compatible donors.Haploidentical transplantation has been certified as a valuable alternative for hematological malignancy patients lacking a well-matched donor, with results comparable matched HLA-identical sibling donors or unrelated donors.The objective of this study is to test the feasibility of haploidentical HSCT for patients with thalassemia major.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with thalassemia major
2. Lacking of a HLA-identical sibling donor or unrelated donor
3. Indication of haploidentical hematopoietic stem cell transplantation
4. No restrictions for transplantation

Exclusion Criteria:

1. Any restriction for transplantation
2. No indication of haploidentical hematopoietic stem cell transplantation

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  2-years overall survival

SECONDARY OUTCOMES:
Disease Free Survival | 2 years
  2-years disease free survival
Engraftment | 30 days
  Myeloid engraftment at day +30
Transplant Related Mortality | 1 year
  Transplant-related mortality by 1 year
Cumulative Incidence of acute Graft Versus Host Disease | 180 days
  Acute graft versus host disease at day +180
Cumulative Incidence of chronic Graft Versus Host Disease | 2 years
  Chronic graft versus host disease by 2 years
Cumulative Incidence of Infectious Complications | 2 years
  Cumulative incidence of bacterial, fungal and viral infections by 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yongrong Lai, MD, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China